CLINICAL TRIAL: NCT05875545
Title: Investigation of the Clinical Effects of Breathing Exercises Combined With Pelvic Floor Exercises in Women With Chronic Pelvic Pain
Brief Title: Effects of Breathing Exercises in Women With Chronic Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 109 (19.10.2022)
Record Dates: First submitted 2023-05-02; First posted 2023-05-25 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2023-04

CONDITIONS: Chronic Pelvic Pain Syndrome; Pelvic Floor; Relaxation; Breathing Exercises; Women
Keywords: Women with Chronic Pelvic Pain; Breathing Exercises; Pelvic Floor Exercises
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing Exercise Group (Active Comparator): Combined breathing and pelvic floor exercises
  Interventions: Other: Breathing Exercises; Other: Pelvic Floor Exercises
- Control Group (Active Comparator): Pelvic floor exercises
  Interventions: Other: Pelvic Floor Exercises

INTERVENTIONS:
Other: Breathing Exercises — Diaphragmatic breathing exercises with a physiotherapist for 8 weeks, two days a week
  Arms: Breathing Exercise Group
Other: Pelvic Floor Exercises — Pelvic floor exercises with a physiotherapist for 8 weeks, two days a week

SUMMARY:
The primary cause of the complex interaction of chronic pelvic pain originates from the visceral organs in the pelvic cavity, and it has been observed that musculoskeletal dysfunctions (such as increased muscle activity in the pelvic floor muscles) are often accompanied by visceral painful stimuli in the pelvic region as a result of shared innervation and visceral-somatic convergence.

This study aims to investigate the effect of breathing exercises combined with pelvic floor exercises on pain, pelvic floor muscle activity, psychological factors, and quality of life in women with chronic pelvic pain.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with chronic pelvic pain (CPA)
* Having pelvic pain for at least 6 months
* 18-45 years old
* Having high resting activity of the pelvic floor (>2 microvolts based on superficial EMG (sEMG) readings)

Exclusion Criteria:

* Having a history of pelvic cancer and/or surgery
* Receiving radiotherapy and/or chemotherapy
* Having a neurological and/or psychiatric pathology
* Have a urinary tract infection
* Menopause
* Presence of current pregnancy status
* History of miscarriage and ectopic pregnancy
* Presence of prolapse
* Being >30 kg/cm2 according to body mass index (BMI)
* Have received treatment for the pelvic area including manual therapy and electrotherapy in the last 6 months
* Having had botulinum toxin injections in the pelvic region in the last 6 months
* Having a communication problem

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women with chronic pelvic pain
Enrollment: 20 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Pelvic Floor Muscle Activity (PFMA) at 8 weeks | at the baseline and end of the 8 weeks (16 sessions)
  PFMA measurement will be performed with the sEMG NeuroTrac MyoPlus Pro (Verity Medical Ltd, UK) device integrated with computer software for digital analysis and report generation.
Change from Baseline Visual Analogue Scale (VAS) at 8 weeks | at the baseline and end of the 8 weeks (16 sessions)
  Pain severity will be evaluated with the VAS.
Change from Baseline McGill Pain Scale- Short Form at 8 weeks | at the baseline and end of the 8 weeks (16 sessions)
  The scale consists of 3 parts. In the first part of the scale, a total of 3 pain scores are obtained: sensory pain score, perceptual pain score and total pain score. In the second part, there were five word groups ranging from "mild pain" to "unbearable pain" to determine the severity of the patient's pain. In the third part, the current pain intensity of the patient was evaluated using a visual comparison scale.

SECONDARY OUTCOMES:
Global Pelvic Floor Disorder Questionnaire | at the baseline and end of the 8 weeks
  Global pelvic floor disorders will be evaluated at baseline and after 8 weeks
Corbin Postural Rating Scale | at the baseline and end of the 8 weeks
  Measuring of posture changes
Pelvic Pain Impact Questionnaire | at the baseline and end of the 8 weeks
  Clinical evaluation of pelvic pain effect
Short Form-36 | at the baseline and end of the 8 weeks
  Evaluation of quality of life
Depression, Anxiety and Stress Scale | at the baseline and end of the 8 weeks
  Evaluation of moods (depression, anxiety and stress)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Saglık Bilimleri University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fall M, Baranowski AP, Elneil S, Engeler D, Hughes J, Messelink EJ, Oberpenning F, de C Williams AC; European Association of Urology. EAU guidelines on chronic pelvic pain. Eur Urol. 2010 Jan;57(1):35-48. doi: 10.1016/j.eururo.2009.08.020. Epub 2009 Aug 31. PMID 19733958
- [Result] Lamvu G, Steege JF. The anatomy and neurophysiology of pelvic pain. J Minim Invasive Gynecol. 2006 Nov-Dec;13(6):516-22. doi: 10.1016/j.jmig.2006.06.021. No abstract available. PMID 17097572
- [Result] Lamvu G, Carrillo J, Witzeman K, Alappattu M. Musculoskeletal Considerations in Female Patients with Chronic Pelvic Pain. Semin Reprod Med. 2018 Mar;36(2):107-115. doi: 10.1055/s-0038-1676085. Epub 2018 Dec 19. PMID 30566976
- [Result] Bradley MH, Rawlins A, Brinker CA. Physical Therapy Treatment of Pelvic Pain. Phys Med Rehabil Clin N Am. 2017 Aug;28(3):589-601. doi: 10.1016/j.pmr.2017.03.009. Epub 2017 May 12. PMID 28676366
- [Result] Klotz SGR MSc, PT, HS, Schon M BSc, PT, Ketels G BA, PT, HE, Lowe B MD, Brunahl CA MD. Physiotherapy management of patients with chronic pelvic pain (CPP): A systematic review. Physiother Theory Pract. 2019 Jun;35(6):516-532. doi: 10.1080/09593985.2018.1455251. Epub 2018 Mar 28. PMID 29589778